CLINICAL TRIAL: NCT02644239
Title: Classic Ketogenic Diet and Modified: Evaluation of the Therapeutic Potential and Impact on the Oxidative Profile, Lipidomic, Inflammatory and Size of Lipoproteins in Children and Adolescents With Refractory Epilepsy
Brief Title: Impact of Ketogenic Diet on Lipoproteins in Refractory Epilepsy
Acronym: Ketonutri
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Patricia Azevedo de Lima, Ph.D. Student, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Faculdade de Saúde Pública USP
Record Dates: First submitted 2015-10-13; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Epilepsy; Cardiovascular Disease; Non-alcoholic Fatty Liver Disease; Quality of Life
MeSH Terms: conditions — Epilepsy; Cardiovascular Diseases; Non-alcoholic Fatty Liver Disease | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group control (Active Comparator): classical ketogenic diet
  Interventions: Dietary Supplement: ketogenic diet
- Group case (Active Comparator): Group case: modified ketogenic diet to reduce at least 20% saturated fat, up> 50% of the acid supply monounsaturated, increasing> 50% polyunsaturated fatty acid content and a lower ratio w6 / w3 at least 50% compared to classic diet used by the control group
  Interventions: Dietary Supplement: ketogenic diet

INTERVENTIONS:
Dietary Supplement: ketogenic diet — Ketogenic diet with high fat (90%)

SUMMARY:
The ketogenic diet is a non-pharmacological treatment prescribed especially for children and indicated in most specialized centers for patients with refractory epilepsy. The composition of the ketogenic diet is based on high-fat, low-carbohydrate, moderate protein content, and the production of ketone bodies is the probable mechanism involved in the control of seizures. The relationship between the treatment of the ketogenic diet and changes in oxidative characteristics, physical and lipid are not well established. Some studies show a significant increase in total cholesterol and triglycerides in children being treated with ketogenic diet, but other studies have shown that changes in lipid profile in the long term do not appear to be significant, beyond the influence of these changes on coronary heart disease are unknown. The studies performed in the last two decades have shown that besides the changes in the lipid profile, oxidative modification of lipoproteins are essential for the initiation and progression of atherosclerosis and physical properties of lipoproteins also appear to be involved in this process, suggesting that the particle size of lipoproteins, through the analysis of subfractions can provide more details of the cardiovascular risk. Thus, this projetct aims to compare the effects of the classical ketogenic diet with the ketogenic diet modified with lower content of saturated fatty acids and a higher content of monounsaturated and polyunsaturated, the oxidative changes of LDL, lipidomic profile, the concentration of antioxidants in production inflammatory cytokines and the subfractions of LDL and HDL in children and adolescents with refractory epilepsy, the clinical effect on controlling epilepsy.

DETAILED DESCRIPTION:
Controlled clinical trial composed of children of adolescents aged 1 to 19 years with refractory epilepsy drug polytherapy (antiepileptic drugs). Children of both sexes are being included. The control group receive the diet classical ketogenic while the case group receive the ketogenic diet modified reduction of at least 20% of the supply of saturated fat and increase> 50% of the acid supply monounsaturated fatty, increase> 50% of acid content polyunsaturated fatty and a lower ratio w6 / w3 at least 50% compared to classical diet used by the control group. Patients are followed in 3 times: baseline, 3 months and 6 months after the intervention.

Exclusion criteria: Children and adolescents who use any type of hormone replacement; Children and adolescents who present diagnosis of diabetes mellitus and hypothyroidism or hyperthyroidism; Children and adolescents with acute illnesses such as heart disease and kidney disease that prevent indication of the DC evaluated by medical history and complete physical examination by the neurologist doctor in charge of the clinic.

Outcome Measures:

a. Characterize the sample as the demographics (gender, age), scioeconomic, quality of life and clinical; B. To assess dietary intake through food records; c. Evaluate the anthropometric profile and classify the nutritional status (Z score of body mass index for age [ZBMI / I]); d. Assess body composition (percentage of fat, lean mass, total body water and phase angle); e. Determine the concentration of cholesterol and triglycerides, lipoproteins (TC, TG, LDL and HDL); f. Determine the concentration of apolipoproteins: APOA-1 and APO-B; g. Detect the concentration of ketone bodies in the plasma (β-hydroxybutyrate); H. Detecting LDL (-) and oxidized LDL in plasma; i. To detect anti-LDL autoantibodies (-) and anti-oxLDL autoantibodies in plasma; j. Determine subfractions HDL, LDL and high LDL particle size; k. To evaluate the concentration of non-esterified fatty acids (NEFAs); l. Assess the concentration of fatty acids in plasma; m. To assess the concentration of substances reactive to thiobarbituric acid (TBARS) in plasma.

n. Determine the concentration of antioxidants in plasma: α-tocopherol, beta-carotene and retinol.

O. Determining the lipidomic plasma profile gathering lipid species in more classes associated with the risk of cardiovascular disease; P. Detecting inflammatory markers: Tumor necrosis factor (TNF-α), interleukin (IL-6) in plasma.

Q. Determine the concentration of hepatic enzymes R. Determine the leptin, adiponectin, ghrelin and resistin S. To evaluate the liver ultrasound and carotid ultrasound

ELIGIBILITY:
Inclusion Criteria: Participate in the study children and adolescents of both sexes with age 1-19 years diagnosed with refractory epilepsy drug polytherapy ( antiepileptic drugs ) and indication of treatment with KD .

-

Exclusion Criteria: Children and adolescents who use any type of hormonal replacement ;

* Children and adolescents who submit diagnosis of diabetes mellitus and hypothyroidism or hyperthyroidism ;
* Children and adolescents showing acute disorders as heart disease and kidney diseases .

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Socioeconomic and clinical profile | average of 3 months
  age, income, disease, parent´s education, use of drugs and supplements, type of seizures, questions about quality of life

SECONDARY OUTCOMES:
Body Mass Index | average of 3 months
  BMI according growth charts
Fat mass | average of 3 months
  Fat mass by impedance bioeletrical
Fat free mass | average of 3 months
  fat free mass by impedance bioeletrical
Phase angle | average of 3 months
  phase angle mass by impedance bioeletrical

OTHER OUTCOMES:
Assessement of food intake | average of 3 months
  Food record applied during 3 days to each time
Ketone bodies | average of 3 months
  Concentration of B-hydroxybutirate in plasma. Determination with kit Ranbut (Randox Laboratories Limited, Reino Unido).
Lipid profile | average of 3 months
  Total cholesterol, LDL, HDL, TG
NEFAS | average of 3 months
  Concentration in plasma. Determination with kit NEFAS(Randox Laboratories Limited, Reino Unido)
LDL oxidized | average of 3 months
  Determination in plasma
Antioxidant | average of 3 months
  Determination of antioxidant concentration in plasma by HPLC
Metabolomic (lipidomic) | average of 3 months
  Determination in plasma by mass spectrometry
Subfractions of Lipoproteins | average of 3 months
  Determination in plasma by Lipoprint
Liver enzymes | average of 3 months
  Concentration of AST, ALT, GGT
Hepatic function | average of 3 months
  Ultrasound liver
Leptin | average of 3 months
  Determination in plasma
Resistin | average of 3 months
  Determination in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Baldini Prudencio, Master, Study Chair — Universidade of Sao Paulo
Locations (1):
- Nagila Raquel Teixeira Damasceno, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Avogaro P, Bon GB, Cazzolato G. Presence of a modified low density lipoprotein in humans. Arteriosclerosis. 1988 Jan-Feb;8(1):79-87. PMID 3341993
- [Background] Avogaro P, Cazzolato G, Bittolo-Bon G. Some questions concerning a small, more electronegative LDL circulating in human plasma. Atherosclerosis. 1991 Nov;91(1-2):163-71. doi: 10.1016/0021-9150(91)90198-c. PMID 1811552
- [Background] Faulin Tdo E, de Sena-Evangelista KC, Pacheco DB, Augusto EM, Abdalla DS. Development of immunoassays for anti-electronegative LDL autoantibodies and immune complexes. Clin Chim Acta. 2012 Jan 18;413(1-2):291-7. doi: 10.1016/j.cca.2011.10.004. Epub 2011 Oct 18. PMID 22037508
- [Background] Fisher RS, Acevedo C, Arzimanoglou A, Bogacz A, Cross JH, Elger CE, Engel J Jr, Forsgren L, French JA, Glynn M, Hesdorffer DC, Lee BI, Mathern GW, Moshe SL, Perucca E, Scheffer IE, Tomson T, Watanabe M, Wiebe S. ILAE official report: a practical clinical definition of epilepsy. Epilepsia. 2014 Apr;55(4):475-82. doi: 10.1111/epi.12550. Epub 2014 Apr 14. PMID 24730690
- [Background] Fisher RS, van Emde Boas W, Blume W, Elger C, Genton P, Lee P, Engel J Jr. Epileptic seizures and epilepsy: definitions proposed by the International League Against Epilepsy (ILAE) and the International Bureau for Epilepsy (IBE). Epilepsia. 2005 Apr;46(4):470-2. doi: 10.1111/j.0013-9580.2005.66104.x. PMID 15816939
- [Background] Freeman JM, Kossoff EH, Hartman AL. The ketogenic diet: one decade later. Pediatrics. 2007 Mar;119(3):535-43. doi: 10.1542/peds.2006-2447. PMID 17332207
- [Background] Kossoff EH, Zupec-Kania BA, Amark PE, Ballaban-Gil KR, Christina Bergqvist AG, Blackford R, Buchhalter JR, Caraballo RH, Helen Cross J, Dahlin MG, Donner EJ, Klepper J, Jehle RS, Kim HD, Christiana Liu YM, Nation J, Nordli DR Jr, Pfeifer HH, Rho JM, Stafstrom CE, Thiele EA, Turner Z, Wirrell EC, Wheless JW, Veggiotti P, Vining EP; Charlie Foundation, Practice Committee of the Child Neurology Society; Practice Committee of the Child Neurology Society; International Ketogenic Diet Study Group. Optimal clinical management of children receiving the ketogenic diet: recommendations of the International Ketogenic Diet Study Group. Epilepsia. 2009 Feb;50(2):304-17. doi: 10.1111/j.1528-1167.2008.01765.x. Epub 2008 Sep 23. PMID 18823325
- [Background] Kwiterovich PO Jr, Vining EP, Pyzik P, Skolasky R Jr, Freeman JM. Effect of a high-fat ketogenic diet on plasma levels of lipids, lipoproteins, and apolipoproteins in children. JAMA. 2003 Aug 20;290(7):912-20. doi: 10.1001/jama.290.7.912. PMID 12928468
- [Background] Lee PR, Kossoff EH. Dietary treatments for epilepsy: management guidelines for the general practitioner. Epilepsy Behav. 2011 Jun;21(2):115-21. doi: 10.1016/j.yebeh.2011.03.008. Epub 2011 Apr 21. PMID 21514240
- [Background] Libby P, Ridker PM, Hansson GK; Leducq Transatlantic Network on Atherothrombosis. Inflammation in atherosclerosis: from pathophysiology to practice. J Am Coll Cardiol. 2009 Dec 1;54(23):2129-38. doi: 10.1016/j.jacc.2009.09.009. PMID 19942084
- [Background] Liu YM, Williams S, Basualdo-Hammond C, Stephens D, Curtis R. A prospective study: growth and nutritional status of children treated with the ketogenic diet. J Am Diet Assoc. 2003 Jun;103(6):707-12. doi: 10.1053/jada.2003.50136. PMID 12778041
- [Background] WHO Multicentre Growth Reference Study Group. WHO Child Growth Standards based on length/height, weight and age. Acta Paediatr Suppl. 2006 Apr;450:76-85. doi: 10.1111/j.1651-2227.2006.tb02378.x. PMID 16817681
- [Background] de Onis M, Onyango AW, Borghi E, Siyam A, Nishida C, Siekmann J. Development of a WHO growth reference for school-aged children and adolescents. Bull World Health Organ. 2007 Sep;85(9):660-7. doi: 10.2471/blt.07.043497. PMID 18026621